CLINICAL TRIAL: NCT01500824
Title: Phase 2 Open-label Single Arm Study Of The Efficacy And Safety Of Crizotinib In East Asian Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) Harboring A Translocation Or Inversion Involving The Anaplastic Lymphoma Kinase (ALK) Gene Locus
Brief Title: A Clinical Study Testing The Safety And Efficacy Of Crizotinib In East Asian Patients With Anaplastic Lymphoma Kinase (ALK) Positive Advanced Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8081027
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Crizotinib; ALK; NSCLC; Non-Small Cell Lung Cancer; Asian
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Crizotinib (Experimental)
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib, 250 mg BID, will be administered orally at approximately the same time each day on a continuous daily dosing schedule

SUMMARY:
This is an open-label multi-center Phase 2 efficacy and safety study of crizotinib in East Asian patients with advanced Non-Squamous NSCLC harboring a translocation or inversion event involving the ALK gene locus who have received only one prior chemotherapy regimen for advanced NSCLC and this regimen must have been platinum-based. Primary objective of this study is to assess the anti-tumor activity and safety profile of crizotinib. Secondary objectives are to evaluate clinical efficacy including median progression-free survival (PFS) and 1-year PFS rate, overall survival (OS), disease control rate (DCR) at 6 and 12 weeks, time to response (TTR), and duration of response (DR).

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of locally advanced or metastatic non-squamous cell carcinoma of the lung
* Positive for translocation or inversion events involving the ALK gene locus
* Patients must have had progressive disease after only one prior chemotherapy regimen. This regimen must have been platinum-based and may have included maintenance therapy.
* Evidence of personally signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.

Exclusion Criteria:

* Current treatment on another therapeutic clinical trial.
* Prior therapy directly targeting ALK.
* Any of the following within the 3 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack.
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade >=2, uncontrolled atrial fibrillation of any grade, or QTc interval >470 msec.
* Pregnancy or breastfeeding.
* Use of drugs or foods that are known potent CYP3A inducers/inhibitors/substrates with narrow therapeutic indices.
* Known HIV infection
* Known interstitial lung disease or interstitial fibrosis
* Other severe acute or chronic medical conditions (including severe gastrointestinal conditions such as diarrhea or ulcer) or psychiatric conditions, or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, and which would, therefore, make the patient inappropriate for entry into this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 33 months

SECONDARY OUTCOMES:
Progression-Free Survival | 33 months
Overall Survival | 33 months
Disease Control Rate | 33 months
Duration of Response | 33 months
Time To Response | 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081027&StudyName=A%20Clinical%20Study%20Testing%20The%20Safety%20And%20Efficacy%20Of%20Crizotinib%20In%20East%20Asian%20Patients%20With%20Anaplastic%20Lymphoma%20Kinase%20%28ALK%29%20Positive